CLINICAL TRIAL: NCT02502851
Title: The Comparison of Strategies to PREPARE Severely CALCified Coronary Lesions Trial (PREPARE-CALC): A Prospective Randomized Controlled Trial of Rotational Atherectomy Versus Cutting/Scoring Balloon in Severely Calcified Coronary Lesions
Brief Title: The Comparison of Strategies to PREPARE Severely CALCified Coronary Lesions Trial (PREPARE-CALC)
Acronym: PREPARE-CALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SK 108 -- 120/14
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Coronary Atherosclerosis Due to Severely Calcified Coronary Lesion
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotational Atherectomy (Active Comparator): Calcified lesion preparation using rotational atherectomy followed by implantation of the ORSIRO sirolimus-eluting stent
  Interventions: Device: Rotational Atherectomy
- Cutting/Scoring Balloon (Active Comparator): Calcified lesion preparation using cutting/scoring balloon followed by implantation of the ORSIRO sirolimus-eluting stent
  Interventions: Device: Cutting/Scoring Balloon

INTERVENTIONS:
Device: Rotational Atherectomy — Calcified lesion preparation using rotational atherectomy before implantation of the Orsiro drug eluting stent
  Arms: Rotational Atherectomy
Device: Cutting/Scoring Balloon — Calcified lesion preparation using cutting/scoring balloons before implantation of the Orsiro drug eluting stent
  Arms: Cutting/Scoring Balloon

SUMMARY:
The primary objective of this study is to evaluate the success of lesion preparation with either rotational atherectomy or cutting/scoring balloons as well as the long term effects of a hybrid sirolimus-eluting stent in an angiographically well-defined group of patients with complex calcified coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical inclusion criteria

   * Age above 18 years and consentable
   * Angiographically proven coronary artery disease
   * Anginal symptoms and/or reproducible ischemia in the target area by ECG, functional stress testing or fractional flow reserve
   * Written informed consent
2. Angiographic inclusion criteria

   * De-novo lesion in a native coronary artery
   * Target reference vessel diameter between 2.25 and 4.0 mm by visual estimation
   * Luminal diameter reduction of 50-100% by visual estimation
   * Severe calcification of the target lesion

Exclusion Criteria:

1. Clinical exclusion criteria

   * Myocardial infarction (within 1 week)
   * Decompensated heart failure
   * Limited long term prognosis due to other conditions
2. Angiographic exclusion criteria

   * Target lesion is in a coronary artery bypass graft
   * Target lesion is an in-stent restenosis
   * Target vessel thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-09; Primary Completion 2018-07 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Strategy Success | Intraprocedural
  The primary endpoint will be 'Strategy Success' defined as successful stent delivery and expansion with attainment of < 20% in-stent residual stenosis of the target lesion in the presence of TIMI 3 flow without crossover or stent failure
In-Stent late lumen loss at 9 months | 9 months
  Co-primary Endpoint: The in-stent late lumen loss at 9 months, defined as the difference between the postprocedure in-stent minimal lumen diameter (MLD) and the in-stent MLD at 9-month followup angiography.

SECONDARY OUTCOMES:
Target vessel failure (TVF) | 9 months, 1 year, 2 years
  Target vessel failure (TVF) defined as a composite of cardiac death, target vessel related myocardial infarction (MI; Q- or non-Q-wave) and clinically driven target vessel revascularization (TVR) at 9 months, 1 and 2 years
In-segment late lumen loss at 9 months | 9 months
  In-segment late lumen loss (stent length + 5 mm on either side) at 9 months
In-segment binary restenosis at 9 months | 9 months
  In-segment binary restenosis (diameter stenosis ≥ 50%) at 9 months
Stent thrombosis at 9 months, 1 and 2 years | 9 months, 1 and 2 years
  Stent thrombosis at 9 months, 1 and 2 years
Peri-procedural MI | within 72 hrs
Procedural duration | Intraproedural
Amount of contrast dye | Intraprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Wahab, MD, Principal Investigator — Segeberger Kliniken GmbH
Locations (1):
- Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Kawaguchi R, Tsurugaya H, Hoshizaki H, Toyama T, Oshima S, Taniguchi K. Impact of lesion calcification on clinical and angiographic outcome after sirolimus-eluting stent implantation in real-world patients. Cardiovasc Revasc Med. 2008 Jan-Mar;9(1):2-8. doi: 10.1016/j.carrev.2007.07.004. PMID 18206630
- [Background] Kuriyama N, Kobayashi Y, Yamaguchi M, Shibata Y. Usefulness of rotational atherectomy in preventing polymer damage of everolimus-eluting stent in calcified coronary artery. JACC Cardiovasc Interv. 2011 May;4(5):588-9. doi: 10.1016/j.jcin.2010.11.017. No abstract available. PMID 21596335
- [Background] Madhavan MV, Tarigopula M, Mintz GS, Maehara A, Stone GW, Genereux P. Coronary artery calcification: pathogenesis and prognostic implications. J Am Coll Cardiol. 2014 May 6;63(17):1703-14. doi: 10.1016/j.jacc.2014.01.017. Epub 2014 Feb 12. PMID 24530667
- [Background] Abdel-Wahab M, Richardt G, Joachim Buttner H, Toelg R, Geist V, Meinertz T, Schofer J, King L, Neumann FJ, Khattab AA. High-speed rotational atherectomy before paclitaxel-eluting stent implantation in complex calcified coronary lesions: the randomized ROTAXUS (Rotational Atherectomy Prior to Taxus Stent Treatment for Complex Native Coronary Artery Disease) trial. JACC Cardiovasc Interv. 2013 Jan;6(1):10-9. doi: 10.1016/j.jcin.2012.07.017. Epub 2012 Dec 19. PMID 23266232
- [Background] Mooney M, Teirstein P, Moses J, Turco M, Reisman M, Waksman R, Saucedo J, Mauri L, Lee D, Gershony G, Mehran R, Carlier S, Lansky A, Leon M. Final Results from the U.S. Multi-Center Trial of the AngioSculpt Scoring Balloon Catheter for the Treatment of Complex Coronary Artery Lesions. Am J Cardiol 2006;98:121.
- [Background] Fonseca A, Costa Jde R Jr, Abizaid A, Feres F, Abizaid AS, Costa R, Staico R, Mattos LA, Sousa AG, Grube E, Sousa JE. Intravascular ultrasound assessment of the novel AngioSculpt scoring balloon catheter for the treatment of complex coronary lesions. J Invasive Cardiol. 2008 Jan;20(1):21-7. PMID 18174614
- [Background] Vaquerizo B, Serra A, Miranda F, Triano JL, Sierra G, Delgado G, Puentes A, Mojal S, Brugera J. Aggressive plaque modification with rotational atherectomy and/or cutting balloon before drug-eluting stent implantation for the treatment of calcified coronary lesions. J Interv Cardiol. 2010 Jun;23(3):240-8. doi: 10.1111/j.1540-8183.2010.00547.x. PMID 20636844
- [Background] Hamon M, Niculescu R, Deleanu D, Dorobantu M, Weissman NJ, Waksman R. Clinical and angiographic experience with a third-generation drug-eluting Orsiro stent in the treatment of single de novo coronary artery lesions (BIOFLOW-I): a prospective, first-in-man study. EuroIntervention. 2013 Jan 22;8(9):1006-11. doi: 10.4244/EIJV8I9A155. PMID 23339805
- [Background] Prati F, Regar E, Mintz GS, Arbustini E, Di Mario C, Jang IK, Akasaka T, Costa M, Guagliumi G, Grube E, Ozaki Y, Pinto F, Serruys PW; Expert's OCT Review Document. Expert review document on methodology, terminology, and clinical applications of optical coherence tomography: physical principles, methodology of image acquisition, and clinical application for assessment of coronary arteries and atherosclerosis. Eur Heart J. 2010 Feb;31(4):401-15. doi: 10.1093/eurheartj/ehp433. Epub 2009 Nov 4. PMID 19892716
- [Background] Kawamori H, Shite J, Shinke T, Otake H, Matsumoto D, Nakagawa M, Nagoshi R, Kozuki A, Hariki H, Inoue T, Osue T, Taniguchi Y, Nishio R, Hiranuma N, Hirata K. Natural consequence of post-intervention stent malapposition, thrombus, tissue prolapse, and dissection assessed by optical coherence tomography at mid-term follow-up. Eur Heart J Cardiovasc Imaging. 2013 Sep;14(9):865-75. doi: 10.1093/ehjci/jes299. Epub 2013 Jan 4. PMID 23291393
- [Derived] Mankerious N, Richardt G, Allali A, Geist V, Kastrati A, El-Mawardy M, Rheude T, Sulimov D, Toelg R, Abdel-Wahab M. Lower revascularization rates after high-speed rotational atherectomy compared to modified balloons in calcified coronary lesions: 5-year outcomes of the randomized PREPARE-CALC trial. Clin Res Cardiol. 2024 Jul;113(7):1051-1059. doi: 10.1007/s00392-024-02434-1. Epub 2024 Mar 14. PMID 38483633
- [Derived] Hemetsberger R, Gori T, Toelg R, Byrne R, Allali A, El-Mawardy M, Rheude T, Weissner M, Sulimov DS, Robinson DR, Richardt G, Abdel-Wahab M. Optical Coherence Tomography Assessment in Patients Treated With Rotational Atherectomy Versus Modified Balloons: PREPARE-CALC OCT. Circ Cardiovasc Interv. 2021 Mar;14(3):e009819. doi: 10.1161/CIRCINTERVENTIONS.120.009819. Epub 2021 Mar 1. PMID 33641372
- [Derived] Abdel-Wahab M, Toelg R, Byrne RA, Geist V, El-Mawardy M, Allali A, Rheude T, Robinson DR, Abdelghani M, Sulimov DS, Kastrati A, Richardt G. High-Speed Rotational Atherectomy Versus Modified Balloons Prior to Drug-Eluting Stent Implantation in Severely Calcified Coronary Lesions. Circ Cardiovasc Interv. 2018 Oct;11(10):e007415. doi: 10.1161/CIRCINTERVENTIONS.118.007415. PMID 30354632